CLINICAL TRIAL: NCT00624390
Title: A Randomized, Masked Patient, Independent Reviewer, Multi-Center Pilot Study to Evaluate the Feasibility of Sepraspray™ Adhesion Barrier in Laparoscopic Myomectomy
Brief Title: Sepraspray™ Laparoscopic Myomectomy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SSPRAY00306
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Laparoscopic Myomectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sepraspray (Experimental): Sepraspray applied directly to both sides of the uterus, Fallopian tubes, and ovaries (or opposing sites if not possible to apply directly). Sepraspray was applied via a sterile cannula at a tissue concentration of approximately 5 mg/cm^2.
  Interventions: Device: Sepraspray
- Control (No Intervention): No anti-adhesion treatment was used.

INTERVENTIONS:
Device: Sepraspray
  Arms: Sepraspray

SUMMARY:
The purpose of this research study is to obtain preliminary data of the safety and effectiveness of Sepraspray in a limited number of patients who are under going a laparoscopic myomectomy. Sepraspray will be applied to the organs in the pelvic cavity following laparoscopic myomectomy. We will compare treatment with Sepraspray as a adhesion prevention barrier after laparoscopic myomectomy versus no adhesion barrier.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a premenopausal women with myomas associated with clinical symptoms deemed suitable for laparoscopic myomectomy and SLL.

Exclusion Criteria:

* Pregnant/lactating women.
* The patient has a history of hypersensitivity to exogenous carboxymethylcellulose products and/or hyaluronic acid.
* The patient's procedure resulted in entry of the endometrial cavity, or entry of the bowel including appendectomy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The safety endpoints will include the type and incidence of AEs, vital signs, wound healing, laboratory examinations, and medication usage. | 30 Days post surgery
Efficacy endpoints are on adhesion formation and will include the success the success criterion for the individual patients as either anterior or posterior uterus free of dense adhesions. | Until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Naperville, Illinois
  - Philadelphia, Pennsylvania
  - Austin, Texas